CLINICAL TRIAL: NCT03353649
Title: Applying Novel Technologies and Methods to Inform the Ontology of Self-Regulation: Binge Eating and Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Russell Alan Poldrack, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5UH2DA041713-02 (NIH); UH2DA041713 (NIH)
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Binge Eating; Smoking, Tobacco; Behavior
MeSH Terms: conditions — Bulimia; Tobacco Smoking; Behavior | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Binge Eating Group (Experimental): (1) exposing subjects to specific stimulus sets relevant to the sample that may promote engagement of appetitive drives (images of highly palatable foods for obese individuals), and (2) exposing them to an instructional manipulation designed to engage self-regulatory processes in the presence of these stimulus sets. Specifically, participants in this sample will be exposed to images of food and control non-food images. In different trials, subjects will be given a "now" cue instructing them to engage with the immediate hedonic properties of the stimulus or a "later" cue instructing them to imagine the long-term consequences of using the stimulus.
  This arm includes fMRI and the now vs. later cue intervention
  Interventions: Behavioral: Now vs. Later Cue; Device: fMRI
- Smoking Group (Experimental): (1) exposing subjects to specific stimulus sets relevant to the sample that may promote engagement of appetitive drives (tobacco-related images or smokers), and (2) exposing them to an instructional manipulation designed to engage self-regulatory processes in the presence of these stimulus sets.
  A similar approach to the Binge Eating sample will be used for the smoking sample using two stimulus sets. Instead of foods and non-food control images, smokers will see smoking-related images and the same control non-food non-smoking images as the Binge Eating sample.
  This Arm includes fMRI and the now vs. later cue intervention
  Interventions: Behavioral: Now vs. Later Cue; Device: fMRI

INTERVENTIONS:
Behavioral: Now vs. Later Cue — As we collect data from all participants, we will include manipulations (or "motivating operations") meant to modulate putative targets within the self-regulation domain in each clinical group - to assess the extent to which we can shift self-regulatory function both in desired and undesired directions. More specifically, subjects will see a "now" cue instructing them to think of immediately using/consuming that stimulus or a "later" cue instruction them to think about the long-term consequences of using/consuming that stimulus. The latter cue is intended to down-regulate desire to use/consume the stimulus, and this down-regulation is measured by a subsequent probe asking subjects the degree to which they want to use/consume that stimulus.
Device: fMRI — Subjects will complete the tasks inside a functional magnetic resonance imaging device, allowing us to measure brain activity that while completing each task.

SUMMARY:
This study aims to examine targets of self-regulatory function among two exemplar populations for which behavior plays a critical role in health outcomes: smokers and individual who binge eat (BED). This is the second phase of a study that aims to identify putative mechanisms of behavior change to develop an overarching "ontology" of self-regulatory processes.

DETAILED DESCRIPTION:
Health risk behavior, including poor diet, physical inactivity, tobacco and other substance use, causes as much as 40% of the illness, suffering, and early death related to chronic diseases. Non-adherence to medical regimens is an important exemplar of the challenges in changing health risk behavior -- and is common, costly (due to increased utilization of healthcare services), and associated with poor patient outcomes. This may be particularly evident among older adults who experience a disproportionate amount of the chronic disease burden in the U.S. Although an array of interventions have been shown to be effective in promoting health behavior change, much of this work has been siloed (focused on one disorder at a time).

Additionally, interventions are typically intended to engage multiple mechanisms of behavior change, but the mechanisms by which they actually work are infrequently systematically examined. Because the need to alter health-related behavior is ubiquitous across medicine, understanding the extent to which the principles of effective health behavior change, and the mechanisms by which they work, are similar or differ across health conditions and settings is a critically important area of scientific inquiry. Improving medical regimen adherence and promoting health behavior change are also crucial issues in the changing healthcare landscape, where quality, value, cost and patient-centered care are central. This line of research may allow for great strides in crafting "precision medicine" approaches for a wide array of populations.

One promising domain of putative behavior change targets is that of self-regulation -- a person's ability to manage cognitive, motivational and emotional resources to act in accordance with his/her long-term goals. In this proposal, the investigators have assembled an outstanding interdisciplinary team to 'scale up' this work to an unprecedented level by examining putative targets of behavior change within the self-regulation mechanism domain across contexts, populations, and assays - in 3 primary levels of analysis: (1) psychological (e.g., constructs such as self-efficacy; emotion regulation; response inhibition), (2) behavioral (e.g., tasks of reward responsiveness; temporal horizon), and (3) biological (structural and functional MRI of key neural circuitry). The investigators will conduct this work with two exemplar populations for which behavior plays a critical role in the course of medical regimen adherence, health, and health outcomes: (1) smokers and (2) binge eaters.

In these groups, the investigators will evaluate the extent to which participants can engage and manipulate putative targets within the self-regulation domain both within and outside of laboratory settings. 50 smokers and 50 obese/overweight persons will participate in a lab study to complete the identified tasks.

The investigators will experimentally modulate engagement of targets (e.g., stimulus set of palatable foods images or tobacco-related images as well as self-regulation interventions).

Subjects will participate in a 30 minute introductory session and a single testing session at Stanford, which will include testing using a subset of self-regulatory tasks from the following list (stop-signal task, conditional motor selective stop signal task, Stroop task, dot pattern expectancy task, attention network task, Columbia card task, task switching, delay discounting task, tower of Hanoi, and emotion regulation task). The order of assessments will be counterbalanced across subjects. Imaging will allow an assessment of the degree to which the neural systems associated with each element in the ontology can be engaged and manipulated in the clinical samples. Imaging will be performed at the Stanford Center for Neurobiological Imaging, which has a research-dedicated 3T GE MRI scanner with all necessary accessories for stimulation and recording. In addition to task-based fMRI, the investigators will collect resting-state fMRI while passively viewing either a blank screen or a movie that may include smoking or food-related stimuli. The proposed sample size of 50 per clinical group will provide sufficient power to detect delta=0.56 between groups, and a correlation of r=0.2 across the aggregated sample.

As the investigators collect data from all participants, they will include manipulations (or "motivating operations") meant to modulate putative targets within the self-regulation domain in each clinical group - to assess the extent to which participants can shift self-regulatory function both in desired and undesired directions. This will be achieved by (1) exposing subjects to specific stimulus sets relevant to the sample that may promote engagement of appetitive drives (images of highly palatable foods for obese individuals, and tobacco-related images or smokers), and (2) exposing them to an instructional manipulation ("now" vs "later" cues that instruct subjects to engage with the immediate hedonistic properties of the stimulus or the long-term consequences of using the stimulus, respectively) designed to engage self-regulatory processes in the presence of these stimulus sets.

ELIGIBILITY:
Inclusion Criteria:

* Understand English sufficiently to provide informed consent
* Right-handed
* Normal or corrected-to-normal vision and no color blindness

Additional Inclusion Criteria for Smoking sample:

* Smoke 5 or more tobacco cigarettes/day for past year
* BMI greater than or equal to 17 and less than 27

Additional Inclusion Criteria for Binge Eating Sample:

* BMI greater than or equal to 27 and less than 45
* Weight limit of 350 lbs
* Non-smoking (defined as no cigarettes in past 12 months-this includes former and never smokers)

Exclusion Criteria:

* Significant medical illness
* History of mental disorder due to a medical condition
* Lifetime history of major psychotic disorders (including schizophrenia and bipolar disorder)
* Current use of any medication for psychiatric reasons (including stimulants and mood stabilizers)

Additional Exclusion criteria for Binge Eating Sample:

* Lost weight in recent past (>10 pounds in past 6 months)
* Currently in a weight-loss program (e.g., Weight Watchers, Jenny Craig)
* Currently on a special diet for a serious health condition

Additional Exclusion Criteria for Smoking Sample:

* Binge eating behavior

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Behavioral Regulation | A single 1.5 hour session for each subject
  Interaction of stimulus class, which is the stimulus of value (smoking stimuli for smokers and palatable foods for binge eaters) vs. neutral control stimuli, with the cue, which is the now vs. later cue. The degree to which subjects can regulate their desire to consume their stimulus of value after a later cue is evidence of successful self regulation.
Regulation of fMRI activation | A single 1.5 hour session for each subject
  Interaction of stimulus class, which is the stimulus of value (smoking stimuli for smokers and palatable foods for binge eaters) vs. neutral control stimuli, with the cue, which is the now vs. later cue. The fMRI activation relating to this interaction is taken as the activation-based neural underpinnings of self-regulation.
Changes in fMRI functional connectivity | A single 1.5 hour session for each subject
  Interaction of stimulus class, which is the stimulus of value (smoking stimuli for smokers and palatable foods for binge eaters) vs. neutral control stimuli, with the cue, which is the now vs. later cue. The fMRI functional connectivity changes relating to this interaction is taken as the connectivity-based neural underpinnings of self-regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford CNI, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon submission of the paper detailing the findings of the research
Access Criteria: All data will be shared openly, with no restrictions on access

REFERENCES:
- [Background] De Jong R, Coles MG, Logan GD. Strategies and mechanisms in nonselective and selective inhibitory motor control. J Exp Psychol Hum Percept Perform. 1995 Jun;21(3):498-511. doi: 10.1037//0096-1523.21.3.498. PMID 7790830
- [Background] Bissett PG, Logan GD. Balancing cognitive demands: control adjustments in the stop-signal paradigm. J Exp Psychol Learn Mem Cogn. 2011 Mar;37(2):392-404. doi: 10.1037/a0021800. PMID 21171806
- [Background] Logan GD, Van Zandt T, Verbruggen F, Wagenmakers EJ. On the ability to inhibit thought and action: general and special theories of an act of control. Psychol Rev. 2014 Jan;121(1):66-95. doi: 10.1037/a0035230. PMID 24490789
- [Background] Hofmann W, Schmeichel BJ, Baddeley AD. Executive functions and self-regulation. Trends Cogn Sci. 2012 Mar;16(3):174-80. doi: 10.1016/j.tics.2012.01.006. Epub 2012 Feb 13. PMID 22336729
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Stroop, J. R. (1935). Studies of interference in serial verbal reactions. Journal of Experimental Psychology, 18, 643-662.
- [Background] Otto AR, Skatova A, Madlon-Kay S, Daw ND. Cognitive control predicts use of model-based reinforcement learning. J Cogn Neurosci. 2015 Feb;27(2):319-33. doi: 10.1162/jocn_a_00709. PMID 25170791
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Casey BJ, Jones RM, Hare TA. The adolescent brain. Ann N Y Acad Sci. 2008 Mar;1124:111-26. doi: 10.1196/annals.1440.010. PMID 18400927
- [Background] Figner B, Mackinlay RJ, Wilkening F, Weber EU. Affective and deliberative processes in risky choice: age differences in risk taking in the Columbia Card Task. J Exp Psychol Learn Mem Cogn. 2009 May;35(3):709-30. doi: 10.1037/a0014983. PMID 19379045
- [Background] Mayr U, Kliegl R. Differential effects of cue changes and task changes on task-set selection costs. J Exp Psychol Learn Mem Cogn. 2003 May;29(3):362-72. doi: 10.1037/0278-7393.29.3.362. PMID 12776747
- [Background] Daugherty, J. R., & Brase, G. L. (2010). Taking time to be healthy: Predicting health behaviors with delay discounting and time perspective. Personality and Individual differences, 48(2), 202-207.
- [Background] Koffarnus MN, Bickel WK. A 5-trial adjusting delay discounting task: accurate discount rates in less than one minute. Exp Clin Psychopharmacol. 2014 Jun;22(3):222-8. doi: 10.1037/a0035973. Epub 2014 Apr 7. PMID 24708144
- [Background] Kirby KN, Marakovic NN. Delay-discounting probabilistic rewards: Rates decrease as amounts increase. Psychon Bull Rev. 1996 Mar;3(1):100-4. doi: 10.3758/BF03210748. PMID 24214810
- [Background] Phillips LH, Wynn VE, McPherson S, Gilhooly KJ. Mental planning and the Tower of London task. Q J Exp Psychol A. 2001 May;54(2):579-97. doi: 10.1080/713755977. PMID 11394063
- [Background] Shallice T. Specific impairments of planning. Philos Trans R Soc Lond B Biol Sci. 1982 Jun 25;298(1089):199-209. doi: 10.1098/rstb.1982.0082. PMID 6125971
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Hu T, Zhang D, Wang J, Mistry R, Ran G, Wang X. Relation between emotion regulation and mental health: a meta-analysis review. Psychol Rep. 2014 Apr;114(2):341-62. doi: 10.2466/03.20.PR0.114k22w4. PMID 24897894
- [Background] Lopresti AL, Hood SD, Drummond PD. A review of lifestyle factors that contribute to important pathways associated with major depression: diet, sleep and exercise. J Affect Disord. 2013 May 15;148(1):12-27. doi: 10.1016/j.jad.2013.01.014. Epub 2013 Feb 14. PMID 23415826

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03353649/Prot_SAP_000.pdf